CLINICAL TRIAL: NCT03574493
Title: Rectal Surgery Evaluation Trial (RESET): Laparotomy vs Laparoscopy vs Robotic vs TaTME Rectal Surgery Matched Parallel Cohort Trial for High Surgical Risk Cancer Patients, With Mid- to Low Rectal Cancer
Brief Title: Rectal Surgery Evaluation Trial (RESET)
Acronym: RESET
Status: Completed | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: PROICM 2018-03 ORE
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Rectal Cancer
Keywords: laparotomy; laparoscopy; low anterior resection; rectal cancer; robot assisted surgery; total mesorectal excision; transanal surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Receptor-Like Protein Tyrosine Phosphatases, Class 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Open laparotomy: A surgical procedure involving a large incision through the abdominal wall to gain access into the abdominal cavity.
  Interventions: Procedure: TME with LAR
- Laparoscopic surgery: A minimally-invasive technique in which operations are performed via small incisions (usually 0.5-1.5 cm) at a location distant to the site of interest.
  Interventions: Procedure: TME with LAR
- Robot-assisted surgery using the da Vinci® Surgical System: A minimally-invasive approach that allows good precision, flexibility, and control.
  Interventions: Procedure: TME with LAR
- Transanal surgery through the anus: Where the protectomy is performed down to up until the Douglas pouch
  Interventions: Procedure: TME with LAR

INTERVENTIONS:
Procedure: TME with LAR — Several surgical techniques are used to perform TME. Dissection using open laparotomy and minimally-invasive laparoscopic or robot-assisted abdominal approaches is performed in a 'top-down' manner, where the instruments are inserted transabdominally and the procedure progresses from splenic flexure/sigmoid colon mobilization to rectal resection. A transanal approach may also be used, a 'bottom-up' procedure where instruments are inserted through the anus to perform rectal resection and TME

SUMMARY:
Total mesorectal excision (TME) is the standard of care for rectal cancer, which can be combined with low anterior resection (LAR) in patients with mid-to-low rectal cancer. The narrow pelvic space and difficulties in obtaining adequate exposure make surgeries technically challenging. Four techniques are used to perform the surgery: open laparotomy, laparoscopy, robot-assisted surgery, and transanal surgery. Comparative data for these techniques is required to provide clinical data on the surgical management of rectal cancers by surgery.

DETAILED DESCRIPTION:
The Rectal Surgery Evaluation Trial will be a prospective, observational, case-matched, four-cohort, multicenter trial designed to study TME with LAR using open laparotomy, laparoscopy, robot-assisted surgery, or transanal surgery in high-surgical-risk patients with mid-to-low, non-metastatic rectal cancer. All surgeries will be performed by surgeons experienced in a technique. Oncologic, morbidity and functional outcomes will be assessed in a composite primary outcome, with success defined as circumferential resection margin ≥1 mm, TME grade III, and minimal postoperative morbidity (absence of Clavien-Dindo grade III-IV complications within 30 days after surgery). Secondary endpoints will include the co-primary endpoints over the long-term (2 years), quality of surgery, quality of life, length of hospital stay, operative time, and rate of unplanned conversions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Rectal adenocarcinoma from middle and lower third (less than 10 cm from the anal verge) with a sphincter saving procedure
3. High risk operative patients (two of these factors as assessed on MRI):

   1. Obese patient with a BMI > 30 (male or female)
   2. Narrow pelvis: inter-tuberous distance < 10 cm
   3. Large tumoral volume with suspicion of close predictive margin (CRM ≤ 1 mm) at diagnosis
   4. Expected coloanal or ultra-low colorectal anastomosis
4. Patients with adequate performance status (Eastern Cooperative Oncology Group Scale score of ≤2)
5. Patient has signed and dated the informed consent before inclusion in the study.

Exclusion Criteria:

1. Patient with a comorbid illness or condition that would preclude the use of surgery.
2. Patients with T4b tumors which impose a pelvectomy
3. Patient requires an abdominal perineal resection (APR)
4. Patients with concurrent or previous invasive pelvic malignant tumors (cervical, uterine, or rectal; excluding the prostate) within 5 years before study enrollment
5. Patient undergoing emergency procedures
6. Planned rectal surgery along with major concomitant procedures (e.g. hepatectomies, other intestinal resections)
7. Metastatic disease
8. Pregnant or suspected pregnancy
9. Patients unwilling to comply with all follow-up study requirements
10. Patient included in another study which impact on the surgical technique or its choice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: high- risk patients with mid-to-low rectal cancer
Sampling Method: Probability Sample
Enrollment: 1098 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of surgical method (success determined by composite of Oncologic, morbidity and functional outcomes) | up to 4 years
  CRM, TME grade III, The absence of clavien dindo grade III-IV complications within 30 days post op

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROUANET, MD, Principal Investigator — ICM Co. Ltd.
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hompes R, Guy R, Jones O, Lindsey I, Mortensen N, Cunningham C. Transanal total mesorectal excision with a side-to-end stapled anastomosis - a video vignette. Colorectal Dis. 2014 Jul;16(7):567. doi: 10.1111/codi.12660. No abstract available. PMID 24801986
- [Background] MacFarlane JK, Ryall RD, Heald RJ. Mesorectal excision for rectal cancer. Lancet. 1993 Feb 20;341(8843):457-60. doi: 10.1016/0140-6736(93)90207-w. PMID 8094488
- [Background] Buchs NC, Nicholson GA, Ris F, Mortensen NJ, Hompes R. Transanal total mesorectal excision: A valid option for rectal cancer? World J Gastroenterol. 2015 Nov 7;21(41):11700-8. doi: 10.3748/wjg.v21.i41.11700. PMID 26556997
- [Background] Sun Z, Kim J, Adam MA, Nussbaum DP, Speicher PJ, Mantyh CR, Migaly J. Minimally Invasive Versus Open Low Anterior Resection: Equivalent Survival in a National Analysis of 14,033 Patients With Rectal Cancer. Ann Surg. 2016 Jun;263(6):1152-8. doi: 10.1097/SLA.0000000000001388. PMID 26501702
- [Background] Vennix S, Pelzers L, Bouvy N, Beets GL, Pierie JP, Wiggers T, Breukink S. Laparoscopic versus open total mesorectal excision for rectal cancer. Cochrane Database Syst Rev. 2014 Apr 15;2014(4):CD005200. doi: 10.1002/14651858.CD005200.pub3. PMID 24737031
- [Background] van der Pas MH, Haglind E, Cuesta MA, Furst A, Lacy AM, Hop WC, Bonjer HJ; COlorectal cancer Laparoscopic or Open Resection II (COLOR II) Study Group. Laparoscopic versus open surgery for rectal cancer (COLOR II): short-term outcomes of a randomised, phase 3 trial. Lancet Oncol. 2013 Mar;14(3):210-8. doi: 10.1016/S1470-2045(13)70016-0. Epub 2013 Feb 6. PMID 23395398
- [Background] Lee SH, Lim S, Kim JH, Lee KY. Robotic versus conventional laparoscopic surgery for rectal cancer: systematic review and meta-analysis. Ann Surg Treat Res. 2015 Oct;89(4):190-201. doi: 10.4174/astr.2015.89.4.190. Epub 2015 Sep 25. PMID 26448918
- [Background] Sun Y, Xu H, Li Z, Han J, Song W, Wang J, Xu Z. Robotic versus laparoscopic low anterior resection for rectal cancer: a meta-analysis. World J Surg Oncol. 2016 Mar 1;14:61. doi: 10.1186/s12957-016-0816-6. PMID 26928124
- [Background] Trastulli S, Farinella E, Cirocchi R, Cavaliere D, Avenia N, Sciannameo F, Gulla N, Noya G, Boselli C. Robotic resection compared with laparoscopic rectal resection for cancer: systematic review and meta-analysis of short-term outcome. Colorectal Dis. 2012 Apr;14(4):e134-56. doi: 10.1111/j.1463-1318.2011.02907.x. PMID 22151033
- [Background] Yang Y, Wang F, Zhang P, Shi C, Zou Y, Qin H, Ma Y. Robot-assisted versus conventional laparoscopic surgery for colorectal disease, focusing on rectal cancer: a meta-analysis. Ann Surg Oncol. 2012 Nov;19(12):3727-36. doi: 10.1245/s10434-012-2429-9. Epub 2012 Jul 3. PMID 22752371
- [Background] Jayne D, Pigazzi A, Marshall H, Croft J, Corrigan N, Copeland J, Quirke P, West N, Rautio T, Thomassen N, Tilney H, Gudgeon M, Bianchi PP, Edlin R, Hulme C, Brown J. Effect of Robotic-Assisted vs Conventional Laparoscopic Surgery on Risk of Conversion to Open Laparotomy Among Patients Undergoing Resection for Rectal Cancer: The ROLARR Randomized Clinical Trial. JAMA. 2017 Oct 24;318(16):1569-1580. doi: 10.1001/jama.2017.7219. PMID 29067426
- [Background] Penna M, Hompes R, Arnold S, Wynn G, Austin R, Warusavitarne J, Moran B, Hanna GB, Mortensen NJ, Tekkis PP; TaTME Registry Collaborative. Transanal Total Mesorectal Excision: International Registry Results of the First 720 Cases. Ann Surg. 2017 Jul;266(1):111-117. doi: 10.1097/SLA.0000000000001948. PMID 27735827
- [Background] Stevenson AR, Solomon MJ, Lumley JW, Hewett P, Clouston AD, Gebski VJ, Davies L, Wilson K, Hague W, Simes J; ALaCaRT Investigators. Effect of Laparoscopic-Assisted Resection vs Open Resection on Pathological Outcomes in Rectal Cancer: The ALaCaRT Randomized Clinical Trial. JAMA. 2015 Oct 6;314(13):1356-63. doi: 10.1001/jama.2015.12009. PMID 26441180
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Baik SH, Kwon HY, Kim JS, Hur H, Sohn SK, Cho CH, Kim H. Robotic versus laparoscopic low anterior resection of rectal cancer: short-term outcome of a prospective comparative study. Ann Surg Oncol. 2009 Jun;16(6):1480-7. doi: 10.1245/s10434-009-0435-3. Epub 2009 Mar 17. PMID 19290486
- [Background] Fleshman J, Branda M, Sargent DJ, Boller AM, George V, Abbas M, Peters WR Jr, Maun D, Chang G, Herline A, Fichera A, Mutch M, Wexner S, Whiteford M, Marks J, Birnbaum E, Margolin D, Larson D, Marcello P, Posner M, Read T, Monson J, Wren SM, Pisters PW, Nelson H. Effect of Laparoscopic-Assisted Resection vs Open Resection of Stage II or III Rectal Cancer on Pathologic Outcomes: The ACOSOG Z6051 Randomized Clinical Trial. JAMA. 2015 Oct 6;314(13):1346-55. doi: 10.1001/jama.2015.10529. PMID 26441179
- [Background] Chessin DB, Enker W, Cohen AM, Paty PB, Weiser MR, Saltz L, Minsky BD, Wong WD, Guillem JG. Complications after preoperative combined modality therapy and radical resection of locally advanced rectal cancer: a 14-year experience from a specialty service. J Am Coll Surg. 2005 Jun;200(6):876-82; discussion 882-4. doi: 10.1016/j.jamcollsurg.2005.02.027. PMID 15922198
- [Background] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S, Quirke P, Couture J, de Metz C, Myint AS, Bessell E, Griffiths G, Thompson LC, Parmar M. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet. 2009 Mar 7;373(9666):811-20. doi: 10.1016/S0140-6736(09)60484-0. PMID 19269519
- [Background] Kang SB, Park JW, Jeong SY, Nam BH, Choi HS, Kim DW, Lim SB, Lee TG, Kim DY, Kim JS, Chang HJ, Lee HS, Kim SY, Jung KH, Hong YS, Kim JH, Sohn DK, Kim DH, Oh JH. Open versus laparoscopic surgery for mid or low rectal cancer after neoadjuvant chemoradiotherapy (COREAN trial): short-term outcomes of an open-label randomised controlled trial. Lancet Oncol. 2010 Jul;11(7):637-45. doi: 10.1016/S1470-2045(10)70131-5. Epub 2010 Jun 16. PMID 20610322
- [Background] D'Agostino RB Jr. Propensity score methods for bias reduction in the comparison of a treatment to a non-randomized control group. Stat Med. 1998 Oct 15;17(19):2265-81. doi: 10.1002/(sici)1097-0258(19981015)17:193.0.co;2-b. PMID 9802183
- [Derived] Rouanet P, Guerrieri M, Lemercier P, Balik E, Cotte E, Spinelli A, Gomez-Ruiz M, Wolthuis A, Bertani E, Dubois A; on behalf the RESET study group. A Prospective European Trial Comparing Laparotomy, Laparoscopy, Robotic-Assisted, and Transanal Total Mesorectal Excision Procedures in High-Risk Patients with Rectal Cancer: The RESET Trial. Ann Surg. 2024 Sep 12. doi: 10.1097/SLA.0000000000006534. Online ahead of print. PMID 39263755
- [Derived] Sgarbura O, Gourgou S, Tosi D, Bakrin N, Bouazza N, Delaine S, De Forges H, Pocard M, Quenet F. MESOTIP: Phase II multicenter randomized trial evaluating the association of PIPAC and systemic chemotherapy vs. systemic chemotherapy alone as 1st-line treatment of malignant peritoneal mesothelioma. Pleura Peritoneum. 2019 Jun 27;4(2):20190010. doi: 10.1515/pp-2019-0010. eCollection 2019 Jun 1. PMID 31417958